CLINICAL TRIAL: NCT06220968
Title: Impact of Glycemic Control on Erectile Function and Penile Doppler in Patients With Erectile Dysfunction
Brief Title: Impact of Glycemic Control on Penile Duplex Results
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mahmoud Abdelradi Khalaf, Resident, Assiut University
Other Study IDs: Penile duplex
Record Dates: First submitted 2023-12-19; First posted 2024-01-24 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Erectile Dysfunction With Diabetes Mellitus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The study aimed at evaluating the impact of glycemic control on the erectile function , penile Doppler, and cavernosal blood NO and glutathione levels among a group of diabetic patients with erectile dysfunction.

DETAILED DESCRIPTION:
Erectile dysfunction (ED) is defined as the inability to achieve or maintain a sufficient erection to engage in sexual intercourse.

Although ED is a benign disorder, it affects physical and psychosocial health and has a significant impact on the quality of life of sufferers and their partners and families. Approximately, 5-20% of men have moderate to severe ED.

Risk factors for ED include age, diabetes, hypertension, obesity, lack of exercise, dyslipidemia, smoking, depression, lower urinary tract symptoms, and pelvic surgery, some of which can be modified. In accordance with the International Society of Impotence Research, ED may be classified into three subtypes: organic (that includes iatrogenic, neurogenic, vasculogenic, and hormonal), psychogenic, and mixed ED. Therefore, a thorough investigation ought to be performed by a multidisciplinary team to avoide misdiagnosis.

In the past, psychogenic cause was considered the most important etiological factor of ED; however, currently, organic factors account for 60-90% of this condition. Endocrinopathies can potentially affect erectile function, most notably hypogonadism, hyperthyroidism, hypothyroidism, and diabetes. The patient's history can raise suspicion for such diagnoses; however, there is significant variability in presentation. To aid in the diagnosis, several screening surveys have been suggested and tested, particularly in the case of hypogonadism. Yet, lack of sensitivity and specificity has led to limited utility. Ultimately, endocrinopathies are evaluated and diagnosed with the use of serum hormonal levels.

Penile erection is a haemodynamic event resulting from a complex interaction between the nervous system and cavernosal tissue (smooth muscle and endothelium). Nitric oxide (NO), synthesized from L-arginine by nitric oxide synthase (NOS), was considered to be the major mediator of corporal smooth muscle cell relaxation.

Lipid peroxidation is thought to be an important biological sequence of oxidative cellular damage. Glutathione (GSH), a substrate of glutathione peroxidase defensive mechanism, is an inhibitor of lipid peroxidation. Thus it is a preventive mechanism for oxidative stress.

Diabetes mellitus (DM) has been associated with erectile dysfunction (ED). The generation of reactive oxygen species (oxidative stress) and the reduction of antioxidant defence in diabetes may play an important role in the aetiology of this complication. Hyperglycaemia may increase the generation of free radicals through glucose oxidation, lipid peroxidation, polyol pathway activation, prostanoid synthesis, non-enzymatic protein glycation, and subsequent oxidative degradation of glycated proteins. Furthermore, exposure of endothelial cells to high glucose leads to augmented production of superoxide anion, which may quench NO. The antioxidant defence mechanisms involve both enzymatic and non-enzymatic strategies. Common antioxidants include vitamins A, C, E, GSH and the enzymes superoxide dismutase, catalase, glutathione peroxidase and reductase. GSH is an electron donor and is able to reduce and to scavenge free radicals; in the reduced form GSH is the most important cell antioxidant. Reduced levels of GSH, due both to a hyperglycaemia-induced increase of free radical production and to a decrease of NADPH levels (like in DM), can impair the endothelial cell functions.

Penile Doppler ultrasound (PDU) study is a diagnostic modality useful in elucidating the cause of ED and the magnitude of its severity. PDU also provides a dynamic, quantifiable and reliable method for evaluation of several structural conditions in the penis. It can also help in detecting fibrotic plaques and calcifications characteristic of Peyronie's disease (PD), defects in the tunica albuginea and variable echogenicity in corpora cavernosa in the case of trauma or features of priapism (differentiating between high and low flow), arteriocavernosal fistulas and high-resistance cavernosal arterial flow in addition to anatomic variations in vasculature. Furthermore, it is suggested that DUS is less time consuming and requires less specialized equipment and facilities than does cavernosometry.

However, despite all these advantages and implications of PDU , it still has some precautions to have a valid result such as experienced physician and good circumstances during examination to alleviate stress and anxiety also type of the used vasoactive substances and their dosing regimen and previous treatment used before the penile imaging that can interfere with the accuracy of the test.

As diabetes mellitus is considered one of the main organic causes of Ed pathophysiology, the investigators are conducting this prospective study to evaluate the impact of glycemic control on erectile function and answer the question of whether diabetic control is a prerequisite before requesting penile duplex for diabetic males with ED in order to have a valid imaging result .

ELIGIBILITY:
Inclusion Criteria:

* Married Male patients diagnosed with erectile dysfunction.
* Age from 30 to 55 years.
* Documented history of DM.
* Regular sexual life with cooperative wife.

Exclusion Criteria:

* Patients with congenital anomalies like hypospadius and curvature.
* History of pelvic or spine surgery.
* Single patient.

  . Thyroid disorders.
* Other sexual disorders.
* Primary ED.
* History of Peyronie's disease or priapism.

Ages: 30 Years to 55 Years | Sex: Male
Age Groups: Adult
Study Population: This prospective observational study will include 100 patients attending our andrology outpatient clinic at Assuit University Hospitals, Egypt, complaining of uncontrolled diabetes mellitus (HBA1C more than 8) and secondary ED for more than 6 months, from October 2023 and over a year. Patients will be included in the study after obtaining a written informed consent and ethical committee approval.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2025-01 (Estimated); Primary Completion 2025-01 (Estimated); Study Completion 2025-03 (Estimated)

PRIMARY OUTCOMES:
Penile doppler ultrasound | Baseline
  penile Doppler and measuring cavernosal blood nitric oxide and glutathione levels to compare penile doppler ultrasound brfore and after glycemic control .
Cavernosal blood nitric oxide | Baseline
  Comparing cavernosal blood nitric oxide brfore and after glycemic control
Cavernosal blood glutathione level | Baseline
  Comparing cavernosal blood glutathione levels brfore and after glycemic control

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed Ab Elshibany, Principal Investigator — Assiut University